CLINICAL TRIAL: NCT04408300
Title: Study of Retinal Vascular Parameters in Patients With Wilson's Disease
Acronym: WILLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APS_2020_5
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Wilson Disease
Keywords: Optical Coherence Tomography; Adaptive optics
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ophthalmological exam (Experimental)
  Interventions: Procedure: Ophthalmological exam

INTERVENTIONS:
Procedure: Ophthalmological exam — Retinophotography, OCT-A (Optical Coherence Tomography- Angiography), OCT-B scan (Optical Coherence Tomography B Scan), Measurement of corrected visual acuity in ETDRS (Early Treatment Diabetic Retinopathy Study), Measurement of intraocular pressure, adaptive optics

SUMMARY:
The rare disease reference center " Wilson disease and other rare copper-related diseases" of the Rothschild Foundation follows a large number of patients with Wilson's with varying degrees of impairment and located at different times of their care.

Many people with Wilson's disease have a characteristic greenish-brown ring, known as Kayser-Fleischer, appearing at the periphery of the cornea due to a deposit of copper at the Descemet membrane. As a general rule, if the patient is compliant with his treatment, the ring usually disappears within a few years, although it may persist in some patients. However, apart from the stage of diagnosis, and the evolution of the ring, ophthalmological examinations are little used for the follow-up of these patients.

The objective of this study is to describe the retinal parameters, in particular vascular with two new retinal imaging technologies (OCT-A :Optical Coherence Tomography-Angiography , Adaptive optics) in patients with Wilson's disease and to correlate them with the parameters of the usual follow-up of these patients (hepatic assessment, exchangeable plasma copper, neurological scores, compliance, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Wilson's disease with Ferenci score ≥4

Exclusion Criteria:

* Neurological or behavioral handicap that does not allow for ophthalmological examinations
* Hepatic decompensation that does not allow for ophthalmological examinations
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Measuring the width of the Kayser-Fleischer ring | Enrollment
  OCT-B scan
Corrected visual acuity measurement | Enrollment
  ETDRS
Intraocular pressure measurement (mmHg) | Enrollment
Measurement of the thickness of the retinal nerve fibers layer (RNFL) | Enrollment
  OCT-B
Measurement of the central avascular zone (in µm2) | Inclusion
  OCT-A
Measurement of the capillary density of the superficial plexus (in%) | Enrollment
  OCT-A
Measurement of the capillary density of the deep plexus (in%) | Enrollment
  OCT-A
Measurement of photoreceptor density (per mm2) | Enrollment
  Adaptive optics
Measurement of wall to lumen ratio (in %) | Enrollment
  Adaptive optics
Measurement of the arterial wall section area (µm²) | Enrollment
  Adaptive optics
Measurement of the diameter of the arterial lumen (µm) | Enrollment
  Adaptive optics

CONTACTS AND LOCATIONS:
Overall Officials: Aurélia POUJOIS, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France